CLINICAL TRIAL: NCT06068010
Title: UVA Protection Factors of SPF 50 and 50+ Face Sunscreens
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP20005-face sunscreens
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Ultraviolet-Induced Change in Normal Skin
Keywords: sunscreen; UVA protection; ISO 24442:2011; photoprotection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to use the International Organization for Standardization (ISO) 24442:2011 in vivo method for assessment of the Ultraviolet A Protection Factor (UVAPF) of topical sunscreen products in healthy adults. The main question it aims to answer is to determine the degree of UVA-protection against UVA radiation.

An area of each subject's skin is exposed to UVA light without any protection and another (different) area is exposed after application of the sunscreen product under test. One further area is exposed after application of a reference UVA sunscreen formulation (S2), which is used to validate the procedure.

DETAILED DESCRIPTION:
The objective of the study conducted in accordance with the Declaration of Helsinki and national regulations regarding human studies is to evaluate the UVA protection factor of the investigational products against UVA, according to the ISO 24442:2011 methodology comparatively to a standard product (Standard S2) in healthy adult subjects.

Standard reference S2 sunscreen formula is used in a study if any test sample has an expected UVAPF of 12 or above. The mean UVAPF for the reference sample S2 is 12,7. The test result of the reference S2 UVAPF must be between 10,7 and 14,7 or the test is invalid and shall be repeated. The reference S2 may be used to validate any product test.

In order to determine the number of subjects, the 95 % confidence interval (CI) shall be taken into account. The 95 % confidence interval should lie within ±17 % of the mean UVAPF, and a minimum of 10 subjects is required.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin phototype: II, III or IV
* colorimetric Individual Typology Angle (ITA°): 20° to 41°
* intact skin on test site

Exclusion Criteria:

* pregnant or lactating women
* subjects using medication with photo-sensitizing potential
* subjects receiving chemotherapy or radiotherapy
* subjects who have had UV exposure on the back area in the four weeks prior to UVAPF testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults meeting the inclusion and exclusion criteria and willing to adhere to the protocol and study procedures
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the protection factor of the investigational product against UVA | from baseline to 24 hours
  The UVAPF test method uses persistent pigment darkening (PPD) responses of the skin as the end point for evaluating transmitted UVA radiation. The test is restricted to the area of the back of selected human subjects. An area of each subject's skin is exposed to UVA light without any protection and another (different) area is exposed after application of the sunscreen product under test. One further area is exposed after application of a reference UVA sunscreen formulation (S2), which is used to validate the procedure.
  To determine the UVAPF, incremental series of UVA exposures are delivered to five or six small sub-sites on the skin to induce darkening responses. These responses are visually assessed for pigment darkness 2 h to 24 h after UVA exposure, by the judgement of a trained evaluator.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Le Floc'h, Study Director — Cosmetique Active International
Locations (6):
- Allergisa, Campinas, Brazil
- France (3):
  - EVIC, Bordeaux
  - Intertek, Paris
  - Eurofins Dermscan France, Villeurbanne
- Eurofins Dermscan Poland, Gdansk, Poland
- CIDP, Bucharest, Romania